CLINICAL TRIAL: NCT02995499
Title: Inter-rater Reliability of the ASA Classification
Acronym: In-ASK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Makridis Georgios, Specialist for Visceral Surgery, Department of General and Visceral Surgery, University Clinic Frankfurt
Other Study IDs: 405/16; U1111-1190-9648 (Other: WHO / UTN)
Record Dates: First submitted 2016-12-11; First posted 2016-12-16 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: ASA PS Klassifikation
Keywords: ASA-PS classification; inter-rater reliability; general surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The ASA-PS classification, a subjective classification system of the patients' preoperative health status, contains a certain problem concerning its interrater reliability. A comparison between anesthesiologic and surgical assessment of the preoperative patient condition has not yet been extensively investigated. The aim of this study is to examine the latter in a prospective, monocentric, observational study.

DETAILED DESCRIPTION:
Included will be prospectively all patients undergoing an operation under anesthesiologic treatment in the one-period-time from the study-beginning at the Department of General and Visceral Surgery of the University Clinic Frankfurt. The ASA-PS classification will be twice conducted and documented during the informed consent process: once by the consulting surgeon and once by the consulting anesthesiologist. The assigned class and the training status of the involved physician are anonymously documented on the study case report form. The pre-, peri- and postoperative patient data, in particular the demographic data (age, height, weight, BMI), comorbidities, type and duration of operation, as well as perioperative complications in a follow-up period of 90 days will be extracted from the electronic patient record. The patient data documentation concludes with a contact and, if necessary, examination of the patient (in hospital or by the family doctor) after the 90th postoperative day. Subsequently two study cooperation partners, a senior surgeon and a senior anesthesiologist, will assign a "recommended"-ASA-PS class to every pseudonymized patient based only on the documented preoperative examination, demographics and comorbidities without insight into the preoperative documented ASA-PS classifications or the postoperative course.

Primary Hypothesis:

The assessments of the preoperative state of health of general-surgical patients by means of the ASA-PS classification carried out independently by members of different disciplines result in a moderate interrater reliability of the latter.

Secondary Hypothesis:

The discrepancy between the abovementioned ASA-PS classification and that recommended by an interdisciplinary committee decreases with increasing professional experience.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing an operation under anesthesiologic treatment in the one-period-time from the study-beginning at the Department of General and Visceral Surgery of the University Clinic Frankfurt.

Exclusion Criteria:

* Patients with ASA-Class 6.
* Patients undergoing surgery more than twice in the same hospital stay (only two evaluations per patient case admitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing an operation under anesthesiologic treatment in the one-period-time from the study-beginning at the Department of General and Visceral Surgery of the University Clinic Frankfurt.
Sampling Method: Non-Probability Sample
Enrollment: 683 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Interrater reliability of the ASA classification | through study completion, an average of 1 year
  Expressed as Krippendorff's alpha and as a Fleiss' kappa

SECONDARY OUTCOMES:
Morbidity rate | 90 days postoperative
  Clavien-Dindo-Klassifikation
Mortality rate | 30 and 90 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Makridis, Dr. med., Principal Investigator — University Clinic Frankfurt; Wolf Otto Bechstein, Prof. Dr., Study Director — University Clinic Frankfurt
Locations (1):
- University Clinic Frankfurt, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No